CLINICAL TRIAL: NCT04680715
Title: Per-Operative Radiotherapy (RPO) by Papillon +TM in Localized Breast Cancer : Faisability and Toxicity Study
Brief Title: Per-Operative Radiotherapy by Papillon +TM in Localized Breast Cancer
Acronym: RPOS+2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/33
Record Dates: First submitted 2020-11-18; First posted 2020-12-23 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Localized Breast Cancer

STUDY DESIGN:
Intervention Model Description: radiotherapy treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Per-Operative Radiotherapy technique by Papillon +TM (Experimental): Per-Operative Radiotherapy (1x20Gy) technique by Papillon +TM
  Interventions: Radiation: Per-Operative Radiotherapy technique by Papillon +TM

INTERVENTIONS:
Radiation: Per-Operative Radiotherapy technique by Papillon +TM — 20Gy Per-Operative Radiotherapy technique by Papillon +TM, on localized breast cancer

SUMMARY:
Phase II study; open recruitment, multicentrique. The aim of this clinical research is to evaluate faisability and toxicity of the per-operative radiotherapy using PAPILLON + TM device for localized breast cancers patients over 65 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient with invasive ductal adenocarcinoma <=2cm, evaluate on all radiological exams;
* Women aged 65 years or older (patients 65 years of age in the year may be included);
* Grade 1 or 2 unifocal adenocarcinoma, all index KI67, positive HR, negative HER2 status;
* T0 or T1, N0 radio-clinic;
* Operable patient with breast volume compatible with conservative surgery;
* Patient with prior malignancy or other concurrent malignancies are eligible, including bilateral breast cancer
* Patients who have been made aware of the information sheet and have given their written signed informed consent;
* Patients benefitting from social health insurance coverage

Exclusion Criteria:

* Age less than 65 years (except if 65 years obtained during the year)
* Patient with an exclusive in situ carcinoma
* Patient with lymphatic invasion / peri-nerve involvement / vascular emboli
* Patient with a lobular adenocarcinoma
* Patient with metastatic disease
* Multifocal tumor
* Patient with grade 3 or N+ disease
* N1 proved by ultrasound guided
* patient unable to express her consent
* Patient deprived placed under the authority of a tutor
* Female patients who are pregnant or breastfeeding
* Vulnerable patient: as defined in article L1121-5 à -8

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
early toxicities occuring until 6 months after performing per-operative radiotherapy | up to 6 months
  pourcentage of patient with toxicities of grade 3 and more (by CTCAE v5.0) related to per-operative radiotherapy and that occured until 6 months after performing

SECONDARY OUTCOMES:
global tolerance of per-operative radiotherapy | up to 5 years
  global safety (assessed by CTCAE V5.0) of per-operative radiotherapy
local disease free survival at 5 years of per-operative radiotherapy | up to 5 years
  To evaluate local disease free survival at 5 years of per-operative radiotherapy
disease free survival at 5 years of per-operative radiotherapy | up to 5 years
  To evaluate disease free survival at 5 years of per-operative radiotherapy
quality of life of patients | up to 6 months
  QLQ-C30 and QLQ BR-23 EORTC questionnaires

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Pôle Santé République, Clermont-Ferrand
  - Centre Antoine Lacassagne, Nice

IPD SHARING:
Plan to Share IPD: No